CLINICAL TRIAL: NCT00622557
Title: General Surgical Outcomes Quality Improvement Database (UH-SOCRATES)
Acronym: SOCRATES
Status: Completed | Type: Observational
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 04-07-18
Record Dates: First submitted 2008-02-11; First posted 2008-02-25 (Estimated); Last update posted 2022-05-12 (Actual); Status verified 2022-05

CONDITIONS: Colon Cancer; Diverticulitis; Colorectal Polyps; Crohn's Disease; Ulcerative Colitis; Rectal Cancer
MeSH Terms: conditions — Colonic Neoplasms; Diverticulitis; Crohn Disease; Colitis, Ulcerative; Rectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Surgical: All patients having surgery procedures

SUMMARY:
A database has been established to track the outcomes of all cases performed in the University Hospitals Department of Surgery in an effort to improve quality of surgical performance and case management.

Specifically, the purpose of the database will be used as a quality improvement tool for analyzing process and outcome measures and to accurately track cases performed by surgeons.

DETAILED DESCRIPTION:
Since the Institute of Medicine report, titled "To Err is Human", there has been an increasing trend to evaluate outcomes in healthcare. While optimal outcomes in delivery of healthcare are something that hospitals and their medical, nursing and administrative staff have always tried to achieve, this has often been attempted without having much information to assess the outcomes that actually occur.

For this reason, programs such as NSQIP (the National Surgical Quality Improvement Project) have been brought from the VA system into private and academic healthcare systems, to sample surgical outcomes and provide hospitals with benchmarks that can be achieved, as well as informing them where they rank in the overall results. Unfortunately, systems such as NSQIP are based on sampling a percentage of cases performed each week, but do not track all cases or all providers. Many cases are therefore not tracked in any way.

Certain centers have now established databases to track their own surgical outcomes. These are usually specific to certain surgical specialties, and provide an opportunity to perform quality improvement. These also have the added value of being useful tools for maintenance of certification and for clinical research.

Primary goals of this study:

We propose to further develop the General Surgical Outcomes Quality Improvement Database(GSOD)-subsequently renamed UH-SOCRATES-which will track all surgical, medical, and radiological encounters occurring at University Hospitals Case Medical Center(UHCMC)as well as at UH's Richmond and Geauga campuses. This database will have several goals:

1. UH-SOCRATES will be used as a quality improvement tool for analyzing process and outcome measures, for example being able to evaluate patients with prolonged length of stay so that cases can be defined and evaluated for specific risk factors or in-hospital events.
2. By using hospital coded CPT codes, UH-SOCRATES will be able to accurately track cases performed by surgeons for maintenance of certification purposes.

All of these goals are related to quality improvement and assessment, and are considered "not human subjects research" under 45 CFR 46. In the future it is hoped that UH-SOCRATES will also be a powerful resource for formal research into surgical outcomes. Future IRB submissions will be submitted for this purpose. This IRB submission therefore only addresses the quality improvement perspective of the UH-SOCRATES.

ELIGIBILITY:
Inclusion Criteria:

* All patients receiving surgical,medical,or radiological services at University Hospitals Case Medical Center,Richmond,or Geauga campuses.

Exclusion Criteria:

* None

Ages: 14 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients receiving surgical, medical, or radiological services at University Hospitals Case Medical Center,Richmond,or Geauga campuses.
Sampling Method: Non-Probability Sample
Enrollment: 200000 (Actual)
Dates: Start 2007-05-01 (Actual); Primary Completion 2017-01-06 (Actual); Study Completion 2017-01-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Conor P. Delaney, MD, PhD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals Case Medical Center, Cleveland, Ohio, United States